CLINICAL TRIAL: NCT05395416
Title: A Phase Ⅱ/Ⅲ Study to Evaluate Efficacy and Safety of Antaitavir Hasophate Capsules in Combination With Yiqibuvir Tablets in Adult Subject With Chronic HCV Infection
Brief Title: Antaitavir Hasophate Capsules Combined With Yiqibuvir Tablets in Treatment Adult Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC74647/HEC110114-Ⅱ/Ⅲ-01
Record Dates: First submitted 2022-05-20; First posted 2022-05-27 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2022-05

CONDITIONS: Chronic HCV Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HEC74647PA+HEC110114 100 mg/200 mg (Experimental): Phase II: HCV GT 1-6 participants were medicated with HEC74647PA Capsules 100 mg or200 mg once daily and HEC110114 tablets 600 mg once daily
  Interventions: Drug: HEC74647PA+HEC110114
- HEC74647PA+HEC110114 (Experimental): Phase III: HCV GT 1-6 participants were medicated with HEC74647PA Capsules 100 mg /200 mg once daily and HEC110114 tablets 600 mg once daily
  Interventions: Drug: HEC74647PA+HEC110114
- Placebo (Placebo Comparator): Phase III: HCV GT 1-6 participants were medicated with HEC74647PA Placebo Capsules once daily and HEC110114 Placebo tablets once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HEC74647PA+HEC110114 — administered orally once daily for 12 weeks
  Other Names: Antaitavir Hasophate+Yiqibuvir
  Arms: HEC74647PA+HEC110114; HEC74647PA+HEC110114 100 mg/200 mg
Drug: Placebo — administered orally once daily for 12 weeks
  Arms: Placebo

SUMMARY:
The safety, tolerability and antiviral activity of Antaitavir Hasophate in Combination With Yiqibuvir in treatment-naive and treatment-experienced patients with chronic hepatitis C virus (HCV) infection

DETAILED DESCRIPTION:
Phase II: Exploring the efficacy and safety of different doses of Antaitavir Hasophate combined with fixed-dose Yiqibuvir in the treatment of adult patients with chronic hepatitis C for 12 weeks, providing a basis for the design and implementation of phase III clinical trials.

Phase III: Confirmation of the efficacy and safety of Antaitavir Hasophate combined with Yiqibuvir in the treatment of adult patients with chronic hepatitis C for 12 weeks, providing a sufficient basis for drug registration and clinical use.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent;
2. Male or female, age≥18 years;
3. Body mass index (BMI)≥18.0 and≤32.0 kg/m2, and Weight≥40 kg;
4. Serological detection of anti-HCV antibodies was positive at screening;
5. HCV RNA≥1×104 IU/mL at Screening;
6. HCV genotype 1~6, mixed genotype or indeterminate assessed at Screening by the Central Laboratory.

Exclusion Criteria:

1. Clinical hepatic decompensation (i.e., ascites, encephalopathy or variceal hemorrhage);
2. Chronic liver disease of a non-HCV etiology (Including but not limited to hemochromatosis, Wilson's disease,alfa-1 antitrypsin deficiency);
3. Significant cardiac disease(Including but not limited to myocardial infarction, bradycardia) ;
4. Psychiatric illness or psychological disease or relevant medical history;
5. Solid organ transplantation;
6. Subjects have any other medical disorder that may interfere with subjects treatment, assessment or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response at 12 weeks after end of treatment (SVR12) | Posttreatment Week 12
  Percentage of subjects with plasma HCV RNA not detected or below the lower limit of quantitation (15 IU/mL)
Type and frequencies of Adverse events | Up to posttreatment week 24
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Percentage of subjects with sustained virologic response 4 and 24 weeks after discontinuation of therapy (SVR4 and SVR24) | Posttreatment Weeks 4 and 24
  SVR4 and SVR24 were defined as HCV RNA < the lower limit of quantitation (LLOQ) at 4 and 24 weeks after stopping study treatment, respectively
Percentage of subjects with virologic failure | Up to posttreatment week 24
  1. On-treatment virologic failure: Breakthrough (confirmed HCV RNA ≥the lower limit of quantitation (LLOQ) after having previously had HCV RNA <the lower limit of quantitation (LLOQ) while on treatment), or Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment);
  2. Virologic relapse: Confirmed HCV RNA ≥the lower limit of quantitation (LLOQ) during the posttreatment period having achieved HCV RNA <the lower limit of quantitation (LLOQ) at last on-treatment visit.

CONTACTS AND LOCATIONS:
Overall Officials: Lai Wei, Doctor, Study Chair — Beijing Tsinghua Changgeng Hospital
Locations (36):
- China (36):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Anhui Provincial Hospital, Hefei, Anwei
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - The 900th Hospital of the Joint Logistics Support Force Hospital, Fuzhou, Fujian
  - Foshan First People's Hospital, Foshan, Guangdong
  - Guangzhou Eighth People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Hainan Provincial People's Hospital, Haikou, Hainan
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Wuhan University People's Hospital, Wuhan, Hebei
  - The Fourth Affiliated Hospital of Harbin Medical University, Haerbin, Heilongjiang
  - Luoyang Central Hospital, Luoyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical College, Xinxiang, Henan
  - Henan Infectious Diseases Hospital, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Zhengzhou People's Hospital, Zhengzhou, Henan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The First Affiliated Hospital of South China, Hengyang, Hunan
  - The First People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - Jiangsu Provincial Hospital, Nanjing, Jiangsu
  - Nanjing Second Hospital, Nanjing, Jiangsu
  - Wuxi No.5 People's Hospital, Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Zhenjiang Third People's Hospital, Zhenjiang, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanyang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Tonghua Central Hospital, Tonghua, Jilin
  - Yanbian University Hospital, Yanbian, Jilin
  - The Sixth People's Hospital Of Shenyang, Shenyang, Liaoning
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Huashan Hospital of the Fudan University, Shanghai, Shanghai Municipality
  - Tianjin Third Central Hospital, Tianjin, Tianjin Municipality
  - Beijing You'an Hospital,Capital Medical University, Beijing